CLINICAL TRIAL: NCT02224443
Title: Effects of Different Doses of Dexmedetomidine on Postoperative Cognitive Dysfunction in Elderly Hypertensive Patients-A Single Center,Randomized, Double-blinded,Controlled Study
Brief Title: Effects of Different Doses of Dexmedetomidine on Postoperative Cognitive Dysfunction in Elderly Hypertensive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Ma Zhengmin, Anaesthetist, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ma sedation
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Dexmedetomidine,postoperative cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Dexmedetomidine; Saline Solution; Midazolam; cisatracurium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A, dexmedetomidine , 0.3µg.kg-1.h-1 (Experimental): Continuous pump infusion dexmedetomidine with loading dose at 0.8µg.kg-1 over 10 minutes,followed Continuous pump infusion dexmedetomidine at 0.3µg.kg-1.h-1 until 30 minutes before end of operation
  Interventions: Drug: dexmedetomidine; Drug: midazolam,fentanyl,etomidate,Cisatracurium besylate; Drug: cisatracurium besylate,propofol,remifentanil,sevoflurane
- Group B,dexmedetomidine , 0.5µg.kg-1.h-1 (Experimental): Continuous pump infusion dexmedetomidine with loading dose at 0.8µg.kg-1 over 10 minutes,followed continuous pump infusion dexmedetomidine at 0.5µg.kg-1.h-1 until 30 minutes before end of operation
  Interventions: Drug: dexmedetomidine; Drug: midazolam,fentanyl,etomidate,Cisatracurium besylate; Drug: cisatracurium besylate,propofol,remifentanil,sevoflurane
- Group C ,normal saline (Placebo Comparator): Normal saline infusion will be given with the same infusion volume as group A and B
  Interventions: Drug: normal saline; Drug: midazolam,fentanyl,etomidate,Cisatracurium besylate; Drug: cisatracurium besylate,propofol,remifentanil,sevoflurane

INTERVENTIONS:
Drug: dexmedetomidine — Experimental: Group A, Continuous pump infusion dexmedetomidine with loading dose at 0.8µg.kg-1 over 10 minutes,followed continuous pump infusion dexmedetomidine at 0.3µg.kg-1.h-1 until 30 minutes before end of operation
  Arms: Group A, dexmedetomidine , 0.3µg.kg-1.h-1
Drug: dexmedetomidine — Group B, Continuous pump infusion dexmedetomidine with loading dose at 0.8µg.kg-1 over 10 minutes,followed continuous pump infusion dexmedetomidine at 0.5µg.kg-1.h-1 until 30 minutes before end of operation
  Arms: Group B,dexmedetomidine , 0.5µg.kg-1.h-1
Drug: normal saline — Group C , Normal saline infusion will be given with the same infusion volume as group A and B
  Arms: Group C ,normal saline
Drug: midazolam,fentanyl,etomidate,Cisatracurium besylate — Anesthesia induction : 0.05 mg.kg-1 midazolam,4~5μg.kg-1 fentanyl,1.0~1.5mg.kg-1etomidate and 0.15 mg.kg-1Cisatracurium besylate
Drug: cisatracurium besylate,propofol,remifentanil,sevoflurane — Maintenance of anesthesia :Continuous pump infusion 0.05~0.1mg.kg-1.h-1cisatracurium besylate,4~8mg.kg-1.h-1propofol,0.1~0.2μg.kg-1.min-1 remifentanil and sevoflurane inhalation with 0.6%~1.0%

SUMMARY:
The purpose of this study is to identify the effects of different doses of dexmedetomidine on postoperative cognitive dysfunction in elderly hypertensive patients

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Elective gastrointestinal surgery
* American Society of Anesthesiologists class II to III
* Aged between 65 and 80 years old
* Weight between 45 and 75 kilogram,Body Mass Index between 19 and 24 kg.m-2
* With primary hypertension reaching or more than 1 year
* Normal cognitive function,mini-mental state examination more than 27

Exclusion Criteria:

* Severe arrhythmia,atrioventricular block and secondary hypertension
* Liver and kidney dysfunction,pulmonary disease,endocrine disease
* Suspected or confirmed difficult airway
* Any disease or pathologic change will interfere study result
* Inability to exchange with serious visual and hearing impairment
* Long term use of sedative-hypnotic drugs and antidepressant drug
* Addicted to alcohol, tobacco or drug
* Neuromuscular disease
* Suspected of malignant hyperthermia
* Allergic to investigational products or with other contraindication
* Participated in other study within 30 days

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to postoperation in cognitive function | One day before operation,third day after operation,sixth day after operaion
  Mini-mental State Examination
Change from baseline to postoperation in recent memory | One day before operation,third day after operation,sixth day after operation
  Rey Auditory Verbal Learning Test
Change from baseline to postoperation in visual space and directional force | One day before operation,third day after operation,sixth day after operaion
  Trail Making Test A,Trail Making Test B
Change from baseline to postoperation in attention | One day before operation,third day after operation,sixth day after operaion
  Digit Span Test
Change from baseline to postoperation in pain scores | One day before operation,third day after operation,sixth day after operation
  Visual analog scales
Change from baseline to postoperation in depression scale | One day before operation,third day after operation,sixth day after operation
  Beck Depression Inventory

SECONDARY OUTCOMES:
The duration of operation | From begining of cutting skin to the end of skin closure,an expected average of 3 hours
The blood volume during the operation | From begining of cutting skin to the end of skin closure,an expected average of 3 hours
The urine volume during operation | From begining of cutting skin to the end of skin closure,an expected average of 3 hours
The dose of drugs used during operation | From begining of cutting skin to the end of skin closure,an expected average of 3 hours
  The dose of ephedrine, urapidil, atropine used during operation